CLINICAL TRIAL: NCT02477553
Title: Describing the Comparative Effectiveness of Colorectal Cancer Screening Tests: The Impact of Quantitative Information
Brief Title: Information With or Without Numbers For Optimizing Reasoning About Medical Decisions
Acronym: INFORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Peter Schwartz, Assistant Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1502774679; CDR-1403-11040 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2015-06-15; First posted 2015-06-23 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Cancer Screening
Keywords: decision aid; cancer screening; colorectal neoplasm; decision making; risk communication; numeracy; health literacy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quantitative (Experimental): Subjects view:
  1. A computer-based presentation regarding colorectal cancer (CRC) and screening for CRC with colonoscopy and stool testing. Includes excerpts from a video from the American Cancer Society.
  2. Computer-based presentation providing quantitative information regarding (a) the lifetime average probability of getting and dying from CRC, (b) the reduction in morbidity and mortality provided by colonoscopy and stool tests, (c) the sensitivity of colonoscopy and stool tests for finding cancer, (d) the false negative values of colonoscopy and stool tests for finding cancer, (e) the risk of heavy bleeding or colon injury from colonoscopy, and (f) the chance of having a positive stool test.
  Interventions: Behavioral: DA - Quantitative
- Verbal (Active Comparator): Subjects view:
  1. A computer-based presentation regarding colorectal cancer (CRC) and screening for CRC with colonoscopy and stool testing. Includes excerpts from a video from the American Cancer Society.
  2. Computer-based presentation providing verbal information regarding (a) the lifetime average probability of getting and dying from CRC, (b) the reduction in morbidity and mortality provided by colonoscopy and stool tests, (c) the sensitivity of colonoscopy and stool tests for finding cancer, (d) the false negative values of colonoscopy and stool tests for finding cancer, (e) the risk of heavy bleeding or colon injury from colonoscopy, and (f) the chance of having a positive stool test.
  Interventions: Behavioral: DA - Verbal

INTERVENTIONS:
Behavioral: DA - Quantitative
  Arms: Quantitative
Behavioral: DA - Verbal
  Arms: Verbal

SUMMARY:
Experts believe that increasing the low uptake of screening for colorectal cancer (CRC) requires educating patients about all approved tests and helping them choose one that fits their preferences. As one motto puts it: "The best test is the one that gets done." Screening tests range from more invasive and very sensitive for polyps and cancer (colonoscopy) to less invasive and less sensitive (e.g., fecal immunochemical testing (FIT)). But it is unclear how best to educate patients about the options and the tradeoffs involved. Some guidelines recommend that decision aids, a promising tool in this area, provide patients with detailed quantitative information, including baseline risk, risk reduction, and chance of negative outcomes. But this sort of "comparative effectiveness" data can confuse patients, especially those with limited mathematical ability. Previous studies have not measured the effect of providing quantitative information to patients with varying levels of ability or interest or asked them whether such data is essential for their decision-making.

The investigators will conduct a clinical trial to determine the impact on patients who view a decision aid (DA) that includes quantitative information versus a DA without such data. The investigators will also seek to determine whether numeracy moderates the effect of quantitative information.

ELIGIBILITY:
Inclusion Criteria:

1. Have not had colonoscopy performed in last 10 years, sigmoidoscopy in last 5 years, or fecal occult blood testing (including FIT) in last 1 year and
2. have a scheduled appointment or due to schedule an appointment with a healthcare practitioner at our performance sites.

Exclusion Criteria:

1. undergoing workup for symptoms consistent with colon cancer, such as weight loss or rectal bleeding
2. have a diagnosis or medical history conferring elevated risk for CRC including polypectomy or colon cancer, inflammatory bowel disease, certain inherited syndromes, or a significant family history of CRC
3. are unable to speak and read English.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Actual)
Dates: Start 2015-06; Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Schwartz, M.D., Ph.D, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from primary care practices between June 2015 and December 2016.
Groups:
- Verbal: Subjects view:
  1. A computer-based presentation regarding colorectal cancer (CRC) and screening for CRC with colonoscopy and stool testing. Includes excerpts from a video from the American Cancer Society.
  2. Computer-based presentation providing verbal information regarding (a) the lifetime average probability of getting and dying from CRC, (b) the reduction in morbidity and mortality provided by colonoscopy and stool tests, (c) the sensitivity of colonoscopy and stool tests for finding cancer, (d) the false negative values of colonoscopy and stool tests for finding cancer, (e) the risk of heavy bleeding or colon injury from colonoscopy, and (f) the chance of having a positive stool test.
  Decision Aid (DA) - Verbal
- Quantitative: Subjects view:
  1. A computer-based presentation regarding colorectal cancer (CRC) and screening for CRC with colonoscopy and stool testing. Includes excerpts from a video from the American Cancer Society.
  2. Computer-based presentation providing quantitative information regarding (a) the lifetime average probability of getting and dying from CRC, (b) the reduction in morbidity and mortality provided by colonoscopy and stool tests, (c) the sensitivity of colonoscopy and stool tests for finding cancer, (d) the false negative values of colonoscopy and stool tests for finding cancer, (e) the risk of heavy bleeding or colon injury from colonoscopy, and (f) the chance of having a positive stool test.
  Decision Aid (DA) - Quantitative
Period: Overall Study
Arm/Group | Verbal | Quantitative
Started | 364 | 364
Completed | 344 | 344
Not Completed | 20 | 20
Not completed — Screening up-to-date | 12 | 13
Not completed — No MD visit | 1 | 1
Not completed — Workup consistent w/CRC | 1 | 1
Not completed — Technical issues with intervention | 2 | 0
Not completed — Elevated risk for CRC | 2 | 2
Not completed — MD advised against screening | 1 | 3
Not completed — patient deceased | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population includes only those participants who completed the study. There were 20 participants in each arm that were withdrawn; these participant's data were not included in the analysis.
Groups:
- Verbal: Subjects view:
  1. A computer-based presentation regarding colorectal cancer (CRC) and screening for CRC with colonoscopy and stool testing. Includes excerpts from a video from the American Cancer Society.
  2. Computer-based presentation providing verbal information regarding (a) the lifetime average probability of getting and dying from CRC, (b) the reduction in morbidity and mortality provided by colonoscopy and stool tests, (c) the sensitivity of colonoscopy and stool tests for finding cancer, (d) the false negative values of colonoscopy and stool tests for finding cancer, (e) the risk of heavy bleeding or colon injury from colonoscopy, and (f) the chance of having a positive stool test.
  DA - Verbal
- Quantitative: Subjects view:
  1. A computer-based presentation regarding colorectal cancer (CRC) and screening for CRC with colonoscopy and stool testing. Includes excerpts from a video from the American Cancer Society.
  2. Computer-based presentation providing quantitative information regarding (a) the lifetime average probability of getting and dying from CRC, (b) the reduction in morbidity and mortality provided by colonoscopy and stool tests, (c) the sensitivity of colonoscopy and stool tests for finding cancer, (d) the false negative values of colonoscopy and stool tests for finding cancer, (e) the risk of heavy bleeding or colon injury from colonoscopy, and (f) the chance of having a positive stool test.
  DA - Quantitative
- Total: Total of all reporting groups
Arm/Group | Verbal | Quantitative | Total
Number analyzed (Participants) | 344 | 344 | 688
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.71 (6.49) | 58.83 (6.66) | 58.77 (6.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 198 | 404
  Male | 138 | 146 | 284
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 5 | 17
  Not Hispanic or Latino | 317 | 329 | 646
  Unknown or Not Reported | 15 | 10 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 98 | 86 | 184
  White | 205 | 232 | 437
  More than one race | 16 | 5 | 21
  Unknown or Not Reported | 20 | 15 | 35
Education [Count of Participants; unit: Participants]
  Less than high school | 25 | 15 | 40
  High school graduate/GED | 75 | 89 | 164
  Some college/technical school/trade school | 92 | 80 | 172
  Associate's degree | 35 | 31 | 66
  Bachelor's degree | 58 | 68 | 126
  Professional or graduate degree | 44 | 51 | 95
  Unknown or Not Reported | 15 | 10 | 25
Relationship [Count of Participants; unit: Participants]
  Single | 71 | 75 | 146
  Married/living with partner | 170 | 168 | 338
  Seperated | 12 | 10 | 22
  Divorced | 61 | 73 | 134
  Widowed | 19 | 8 | 27
  Unknown or Not Reported | 11 | 10 | 21
Employed? [Count of Participants; unit: Participants]
  Yes | 158 | 188 | 346
  No | 170 | 146 | 316
  Unknown or Not Reported | 16 | 10 | 26
Health Insurance? [Count of Participants; unit: Participants]
  Yes | 315 | 317 | 632
  No | 13 | 17 | 30
  Unknown or Not Reported | 16 | 10 | 26
Insurance Lapse over past 12 months? [Count of Participants; unit: Participants]
  Yes | 51 | 46 | 97
  No | 278 | 286 | 564
  Unknown or Not Reported | 15 | 12 | 27
Self-reported health status at baseline [Count of Participants; unit: Participants]
  Excellent | 23 | 33 | 56
  Very good | 87 | 111 | 198
  Good | 144 | 133 | 277
  Fair | 63 | 51 | 114
  Poor | 11 | 6 | 17
  Unknown or Not Reported | 16 | 10 | 26
Income Level (yearly) [Count of Participants; unit: Participants]
  Less than $20,000 | 95 | 80 | 175
  $20,000 - $39,999 | 59 | 73 | 132
  $40,000 - $59,000 | 37 | 40 | 77
  $60,000 - $99,999 | 67 | 63 | 130
  More than $100,000 | 47 | 56 | 103
  Unknown or Not Reported | 39 | 32 | 71
Income Level Subjective [Count of Participants; unit: Participants]
  Are comfortable | 129 | 145 | 274
  Have just enough to make ends meet | 117 | 125 | 242
  Do not have enough to make ends meet | 80 | 59 | 139
  Unknown or Not Reported | 18 | 15 | 33

OUTCOME MEASURES:

1. Primary Outcome: Colorectal Cancer (CRC) Screening Completion
Description: Completion of colonoscopy, fecal immunochemical testing (FIT), or other CRC screening test within 6 months of enrollment, based on documentation in the participants' electronic health record. If a patient completed both screening tests and the colonoscopy was a follow-up to a positive FIT, they were considered having completed a FIT only. If the FIT was negative and the patient still had a colonoscopy, they were considered to have completed both tests.
Time Frame: 6 months post intervention
Population: All participants who agreed to having their electronic health record (EHR) checked by the researchers. There were 12 participants in the Verbal arm and 4 participants in the Quantitative arm who would not agree for their EHRs to be checked by the researchers; therefore, assessment of uptake was not performed with those participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Verbal | Quantitative
Number analyzed (Participants) | 332 | 340
Participants | 99 | 99

2. Primary Outcome: Colorectal Cancer (CRC) Screening Intention: Change From Baseline to Post-intervention
Description: Multiple choice question assessing subject's intention in getting a CRC screening test in the next 6 months. The response options were: 5=Definitely, 4=Probably, 3=May or may not, 2=Probably not, and 1=Definitely not. Higher positive change means CRC screening intention increased. Increased intention to be screened is a better outcome.
Time Frame: 1 day (baseline [before viewing decision aid] and post-intervention [immediately after viewing decision aid])
Population: All participants with both baseline and post-intervention responses to CRC screening intent items. There were 2 participants in each arm who did not respond to at least one of the intent items.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Verbal | Quantitative
Number analyzed (Participants) | 342 | 342
units on a scale | 0.37 (0.84) | 0.47 (0.84)

3. Secondary Outcome: Perceived Risk of Colorectal Cancer (CRC): Change From Baseline to Post-intervention
Description: Multiple choice questions assessing subject's perception of how likely they are to get colon cancer in the next 5 years, in the next 10 years, and sometime during their lifetime. Each had response options: 4=very likely, 3=somewhat likely, 2=somewhat unlikely, and 1=very unlikely. The mean of the 3 questions was calculated (each combined score has a range of 1 to 4) at baseline and post-intervention and then change from baseline was calculated using the mean at post-intervention minus the mean at baseline. The range for change could be from -3 to 3 with higher values meaning an increase in perceived risk which is a better outcome.
Time Frame: 1 day (baseline [before viewing decision aid] and post-intervention [immediately after viewing decision aid])
Population: All participants with baseline (T0) and post-intervention (T1) perceived risk items. Missing responses were not used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Verbal | Quantitative
Number analyzed (Participants) | 333 | 336
units on a scale | -0.08 (0.70) | 0.08 (0.81)

4. Secondary Outcome: Perceived Benefits of Colorectal Cancer Screening With Fecal Immunochemical Test (FIT) and Colonoscopy: Change From Baseline to Post-intervention
Description: Assessed separately for colonoscopy (4 questions) and FIT (4 questions), using items drawn from validated scales for measuring benefits and self-efficacy of colonoscopy and FIT. All items had Likert-type response options where 5=strongly agree to 1=strongly disagree. Mean values were calculated within each set of questions (each combined score has a range of 1 to 5) at baseline and post-intervention and then change from baseline was calculated using the mean at post-intervention minus the mean at baseline. The range for change could be -4 to 4 with higher values meaning perceived benefits increased which is a better outcome.
Time Frame: 1 day (baseline [before viewing decision aid] and post-intervention [immediately after viewing decision aid])
Population: Participants who completed both the baseline and post-intervention benefit questions. For colonoscopy, it was 324 in Verbal and 332 in Quantitative. For FIT, it was 320 in Verbal and 330 in Quantitative.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Verbal | Quantitative
Number analyzed (Participants) | 324 | 332
units on a scale
  Colonoscopy Benefits | 0.44 (0.62) | 0.47 (0.62)
  FIT Benefits: number analyzed (Participants) | 320 | 330
  FIT Benefits | 0.44 (0.76) | 0.52 (0.73)

5. Secondary Outcome: Perceived Barriers to Colorectal Cancer Screening With Fecal Immunochemical Test (FIT) or Colonoscopy: Change From Baseline to Post-intervention
Description: Assessed separately for colonoscopy (11 questions) and FIT (9 questions), using items drawn from validated scales for measuring barriers and self-efficacy of colonoscopy and FIT. All items had Likert-type response options where 5=strongly agree to 1=strongly disagree. Mean values were calculated within each set of questions (each combined score has a range of 1 to 5) at baseline and post-intervention and then change from baseline was calculated using the mean at post-intervention minus the mean at baseline. The range for change could be -4 to 4 with lower values meaning perceived barriers decreased which is a better outcome.
Time Frame: 1 day (baseline [before viewing decision aid] and post-intervention [immediately after viewing decision aid])
Population: Participants who completed both the baseline and post-intervention barrier questions. For colonoscopy, it was 322 in Verbal and 330 in Quantitative. For FIT, it was 321 in Verbal and 327 in Quantitative.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Verbal | Quantitative
Number analyzed (Participants) | 322 | 330
units on a scale
  Colonoscopy Barriers | -0.18 (0.47) | -0.13 (0.45)
  FIT Barriers: number analyzed (Participants) | 321 | 327
  FIT Barriers | -0.18 (0.55) | -0.21 (0.54)

6. Secondary Outcome: Knowledge of Colorectal Cancer (CRC) and Colorectal Cancer Screening: Change in Number of Correct Answers From Baseline to Post-intervention
Description: Qualitative knowledge is assessed with five multiple choice and five true/false questions regarding general information (including risk factors, screening test options, and test frequency) of CRC and CRC screening. Knowledge scores were derived by summing correct responses to the 10 individual knowledge questions (range, 0-10), and change from baseline was calculated using the knowledge score at post-intervention minus the knowledge score at baseline. The range for change could be 0 to 10 with higher values meaning an increase in knowledge which is a better outcome.
Time Frame: 1 day (baseline [before viewing decision aid] and post-intervention [immediately after viewing decision aid])
Population: All participants who completed at least 7 knowledge questions at both baseline (T0) and post-intervention (T1).
Measure: Mean (Standard Deviation); unit: correct answers
Arm/Group | Verbal | Quantitative
Number analyzed (Participants) | 342 | 342
correct answers | 3.13 (2.99) | 3.66 (2.82)

7. Secondary Outcome: Decision Conflict: Change in Conflict From Baseline to Post-intervention
Description: Decision conflict is assessed using the16-item Decision Conflict Scale. Scores will range from 0 (low decision conflict) to 100 (high decision conflict). Negative change means decision conflict decreased. A decrease in decision conflict is a better outcome.
Time Frame: 1 day (baseline [before viewing decision aid] and post-intervention [immediately after viewing decision aid])
Population: All participants with at least 11 responses to the 16-item Decision Conflict Scale at both baseline (T0) and post-intervention (T1).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Verbal | Quantitative
Number analyzed (Participants) | 316 | 326
units on a scale | -19.3 (17.77) | -22.0 (19.25)

8. Secondary Outcome: Number of Patients With High and Low Subjective Numeracy
Description: Subjective numeracy was determined using the Subjective Numeracy Scale (SNS), a validated instrument that involves 8 Likert-type questions regarding the participant's preference for or dislike of numeric information and their perception of their ability to understand it. Each item has a six-point response option from 1-6. The higher the number, the higher the subjective numeracy. All participants were divided into two groups: above (high numeracy) and below (low numeracy) the median for their total subjective numeracy score.
Time Frame: 1 day
Population: Subjects who completed the Subjective Numeracy Scale.
Measure: Count of Participants; unit: Participants
Arm/Group | Verbal | Quantitative
Number analyzed (Participants) | 336 | 337
Participants
  Low Subjective Numeracy | 172 | 160
  High Subjective Numercy | 164 | 177

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Quantitative | Verbal
All-Cause Mortality (participants affected / at risk) | 0/364 | 0/364
Serious Adverse Events (participants affected / at risk) | 0/364 | 0/364
Other Adverse Events (participants affected / at risk) | 0/364 | 0/364

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT02477553/Prot_SAP_000.pdf